CLINICAL TRIAL: NCT01303588
Title: Yoga and Qigong for Elderly Patients With Chronic Low Back Pain
Acronym: YQ-LBP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YQ-LBP
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Low Back Pain
Keywords: elderly patients
MeSH Terms: conditions — Low Back Pain | interventions — Yoga; Qigong

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Waiting Group (No Intervention)
- Qigong (Active Comparator)
  Interventions: Behavioral: Qigong
- Yoga (Active Comparator)
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — 24 group training sessions Yoga, 2 training sessions per week, 45 min duration , over 3 months
  Arms: Yoga
Behavioral: Qigong — 12 group training sessions Qigong, 1 training per week, 90 min duration , over 3 months
  Arms: Qigong

SUMMARY:
The objective of this study is to evaluate whether yoga or qigong therapy is effective in treating low back pain in elderly patients compared to no therapy (waiting list control). The secondary aim is to compare yoga and qigong.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 65 years of age
* Chronic low back pain since 6 months at least
* Functional Rating Index (FRI) ≥ 2 last 7 days
* Informed consent form signed

Exclusion Criteria:

* Disc prolapse with acute neurological symptoms
* Previous spinal operations
* Severe organic or psychiatric disease conditions, not allowing to participate in the trial
* Use of opioids
* Drug- and alcohol-addiction
* Participation in another clinical trial within the last 6 months
* Participation in yoga or qigong training within the last 12 months
* Planned physical therapy within study duration

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 176 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Functional rating Index (FRI) | 3 months

SECONDARY OUTCOMES:
Functional Rating Index | 6 months
Visual Analogue Scale | 3, 6 months
FFb-HR | 3, 6 months
Pain medication | 6 months
Falls | 6 months
Tinetti Test | 3, 6 months
SF 36 | 3, 6 months
Geriatric Depression Scale | 3, 6 months
Adverse events | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Berlin, Institute for Social Medicine, Epidemiology, Health Economics, Berlin, State of Berlin, Germany